CLINICAL TRIAL: NCT06455592
Title: Effect of Practicing Adapted Physical Activity (APA) on Sleep Quality in Children From 5 Years of Age and Adolescents up to 16 Years of Age Undergoing Treatment for a Hematologic Malignancy.
Brief Title: Effect of APA on Sleep Quality in Children With Cancer From 5 to 16 Years
Acronym: APANYX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AOI 2022 LABRAISE; 2023-A02575-40 (Other: 2023-A02575-40)
Record Dates: First submitted 2024-05-31; First posted 2024-06-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Child, Only; Blood Cancer; Adapted Physical Activity; Sleep
Keywords: child; blood cancer; adapted physical activity; sleep; hospital and home
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: experimental, randomized, cross-over, single-center therapeutic trial, controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard (Active Comparator): practice only once adapted physical activity in hospital and at home during four days
  Interventions: Other: control arm
- daily adapted physical activity (Experimental): practice adapted physical activity daily in hospital and at home during four days
  Interventions: Behavioral: practice adapted physical activity

INTERVENTIONS:
Behavioral: practice adapted physical activity — practice daily adapted physical activity during 4 days
  Arms: daily adapted physical activity
Other: control arm — practice once adapted physical activity during 4 days
  Arms: standard

SUMMARY:
Main objective :

Evaluate the effect of adapted physical activity on the sleep of children with cancer from 5 to 16

Hypothesis :

Practice daily adapted physical activity improve the sleep of the 5 to 16 children with cancer

DETAILED DESCRIPTION:
Medical process are leading to an increase in the survival of children/adolescents undergoing treatment for blood cancer. Caregivers need to focus on optimizing these patients' quality of life during and after the disease. Sleep is essential to their development. Sleep disorders are symptoms reported by patients. They have a negative impact on their quality of life. Adapted physical activity sessions are offered in pediatric oncology departments, but sedentary behavior persists. The hypothesis is that the daily practice of adapted physical activity will improve sleep in patients treated for blood cancer.

This is a randomized, cross-over, open-label, two-armed parallel, unique center therapeutic trial comparing the effect of practice adapted physical activity only once during four days (conventional strategy) versus practice adapted physical activity each day during four days (experimental strategy) on the sleep of the children with blood cancer from 5 to 16 at the hospital in Clermont-Ferrand and at home.

The study will last four weeks with a wash-out week after 2 weeks. The outcomes are described later. The nurse informs and obtains the consent of the child and his parents. After statistical analysis of these two arms, it will be possible to determine the value of practice daily adapted physical activity on the sleep of children with blood cancer from 5 to 16 at the hospital and at home.

ELIGIBILITY:
Inclusion Criteria:

* Children from 5 to 16 with haematological cancer undergoing treatment
* Subjects and their parents who were informed about the study and gave informed consent.
* Enrollment in the Social Security system

Exclusion Criteria:

* Children on high-dose corticosteroids
* Children under anxiolytic treatment
* Children with sleep disorders (sleep apnea)
* Children taking melatonin or sleeping pills
* Contraindication to adapted physical activity
* Refusal to participate on the part of the participant or his/her parents
* Holders of parental authority under curatorship, guardianship, safeguard of justice
* Pregnant or breast-feeding teenagers

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Quality of sleep | the morning and the evening, from the morning of the first day to the morning of the fourth day, during the 2 sessions of 2 cycles, each cycle is 4 days
  daily calendar with information about child's sleep complete by parents

SECONDARY OUTCOMES:
Number of sleep's hour and night awakenings | Each night from the bedtime to the wake up time, from the bedtime of the first day to the wake up time of the fourth day, during the 2 sessions of 2 cycles, each cycle is 4 days
  wear a sleep recorder during the night
rate of daily human physical activity in met/day | from the morning of the first day to the morning of the fourth day, during the 2 sessions of 2 cycles, each cycle is 4 days
  wear a wearable device allday and night long
children quality of life | the morning the fourth day, during the 2 sessions of 2 cycles, each cycle is 4 days
  parent-completed questionnaire
chair stand-up test | the morning of the first day and the morning of the fourth day, during the 2 sessions of 2 cycles, each cycle is 4 days
  maximum sit-up and stand-up from a chair during one minute
vigilance status description | at 10am, 2pm and 6pm from the first day to the third day and only at 10am the fourth day, during the 2 sessions of 2 cycles, each cycle is 4 days
  parent-completed questionnaire
children's pain self evaluation | at 8am and 6pm from the first day to the third day and only at 8am the fourth day, during the 2 sessions of 2 cycles, each cycle is 4 days
  self evaluation of children's pain with the visial analog scale in vertical position quote from 0 to 10, 10=worst score
fatigue status | at 10am, 2pm and 6pm from the first day to the third day and only at 10am the fourth day, during the 2 sessions of 2 cycles, each cycle is 4 days
  parent-completed questionnaire
inflammation markers | the morning, from the first and the fourth day, during the 2 sessions of 2 cycles, each cycle is 4 days
  C reactive protein and IL6 from daily blood test

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle LABRAISE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No